CLINICAL TRIAL: NCT06870552
Title: Core Semantic Systems of the Human Brain
Brief Title: Core Semantic Systems TMS
Acronym: CSST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Rutvik H. Desai, Professor, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00098791; R01DC017162 (NIH)
Record Dates: First submitted 2024-09-23; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Lexical Access in Neurotypicals
Keywords: semantic processing; time course; lexical access; anterior temporal lobe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TMS (Experimental)
  Interventions: Device: Single-pulse TMS

INTERVENTIONS:
Device: Single-pulse TMS — A single pulse TMS is delivered at different time points when processing words or numbers.

SUMMARY:
This study examines the time course of activation of the left anterior temporal lobe (ATL) during lexical processing using Transcranial Magnetic Stimulation (TMS).

DETAILED DESCRIPTION:
This study investigates the activation time of the anterior temporal lobe (ATL) region during lexical processing. Participants will perform three tasks: lexical decision, semantic decision (divided into noun and verb semantic decision), and number judgment.

Lexical Decision Task: Participants will be shown words and pseudowords (e.g., excaid). Participants have to decide if the presented stimulus is a real word or a pseudoword.

Semantic Decision Task: Participants will determine if the stimulus word refers to an action or an object that can be manipulated using the hand or arm.

Half of the stimuli will be nouns, constituting the first semantic decision task with objects, and the other half will be verbs, constituting the second semantic decision task with actions.

Number Judgment Task: Participants will decide if a presented number was divisible by four (e.g., 64) or not (e.g., 69). The stimuli will include numbers with either two or three digits.

For each task, we will collect accuracy and reaction time (RT) data. The primary analyses concern the RTs, but accuracies will also be examined in secondary analyses.

A single pulse TMS will be applied at three different time points: -100 ms, 150 ms, and 400 ms after the onset of the stimulus item. A Magstim BiStim² stimulator with a figure-8 coil will be used. The resting motor threshold (RMT) will be defined as the minimum intensity required to stimulate the motor cortex, eliciting a contraction of the abductor pollicis brevis in at least 5 out of 10 trials. The coil will be positioned at a 45-degree angle along the parasagittal line on the presumed motor cortex area for the APB muscle and adjusted in different directions to find the optimal motor hotspot. Intensity will be between 100% and 120% of resting motor threshold as tolerated by the participant.

The effect of TMS on the response time (RT) at different time points will be examined. TMS will be applied at the left anterior middle temporal gyrus at 10 mm posterior to the tip of the temporal pole. A structural MRI scan will be collected prior to the TMS, which will be used in localizing The target spot. A BrainSight neuronavigation system will be used, with the MRI scan collected before, to localize the target location on the scalp. The tasks will last approximately 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be within the ages of 18 to 40
* Native speakers of English

Exclusion Criteria:

* Potential participants with a clinically reported history of dementia, alcohol abuse, psychiatric or neurological disorders, traumatic brain injury, or extensive vision or hearing problems that prevents them from performing the tasks
* Contraindication to TMS, determined by a standard TMS screening form
* Contraindication to MRI, determined by a standard MRI screening form
* Left handed participants

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Mean reaction time changes in lexical decision from TMS at 150 ms | Through study completion, an average of 1 year.
  An interaction between time point (-100, 150) and task (lexical decision, number judgment) RT at the group level (one tailed).
  (LD_150 - LD_-100) - (NJ_150 - NJ_-100).

SECONDARY OUTCOMES:
Mean reaction time changes in semantic decision from TMS at 150 ms | Through study completion, an average of 1 year.
  An interaction between time point (-100, 150) and task (semantic decision, number judgment) RT at the group level (one tailed).
  (SD_150 - SD_-100) - (NJ_150 - NJ_-100).

OTHER OUTCOMES:
Mean reaction time changes in lexical decision from TMS | Through study completion, an average of 1 year.
  LD RT at -100 ms will be lower than LD RT at 150 ms.
Mean reaction time changes in semantic decision from TMS | Through study completion, an average of 1 year.
  Sematic decision RT at -100 will be lower than RT at 150 ms.
Mean reaction time changes in lexical decision from TMS at 400 ms | Through study completion, an average of 1 year.
  An interaction between time point (-100, 400) and task (lexical decision, number judgment) RT at the group level (one tailed).
  (LD_400 - LD_-100) - (NJ_400 - NJ_-100).
Mean reaction time changes in semantic decision from TMS at 400 ms | Through study completion, an average of 1 year.
  An interaction between time point (-100, 400) and task (semantic decision, number judgment) RT at the group level (one tailed). These effects will be examined separately for nouns and verbs as well.
  (SD_400 - SD_-100) - (NJ_400 - NJ_-100).
Mean reaction time changes in noun semantic decision from TMS at 150 ms | Through study completion, an average of 1 year.
  An interaction between time point (-100, 150) and task (semantic decision of nouns, number judgment) RT at the group level (one tailed). (SD_noun_150 - SD_noun_-100) - (NJ_150 - NJ_-100).
Mean reaction time changes in verb semantic decision from TMS at 150 ms | Through study completion, an average of 1 year.
  An interaction between time point (-100, 150) and task (semantic decision of verbs, number judgment) RT at the group level (one tailed). (SD_verb_150 - SD_verb_-100) - (NJ_150 - NJ_-100).

CONTACTS AND LOCATIONS:
Locations (1):
- Prisma Health Richland, Columbia, South Carolina, United States